CLINICAL TRIAL: NCT02076360
Title: Impact of Preoperative Patient Education Video on Patient Preparedness After Sacrocolpopexy: A Single Blind Randomized Controlled Trial
Brief Title: RCT: Impact of Preop Video on Patient Preparedness for Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00013617
Record Dates: First submitted 2013-09-20; First posted 2014-03-03 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2016-05

CONDITIONS: Prolapse
Keywords: Preoperative counseling; Patient satisfaction; Prolapse; Sacrocolpopexy
MeSH Terms: conditions — Prolapse; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preop Video (Experimental): This arm will watch an instructional video in addition to their normal preoperative visit with the physician.
  Interventions: Behavioral: Preoperative Video
- No video (No Intervention): This arm will receive only the normal preoperative visit with the physician without the additional video

INTERVENTIONS:
Behavioral: Preoperative Video — Patients will watch preoperative instructional video
  Arms: Preop Video

SUMMARY:
This is a single-blind, randomized (1:1 allocation), stratified, single-parallel clinical trial at one institution evaluating the use of a preoperative patient education video as an adjunct to preoperative counseling on patient-centered outcomes.

The aim of this study is to determine the impact of a preoperative patient educational video as an adjunct to the routine preoperative visit on patients' preparedness for surgery, perception of time spent with their healthcare team, and ultimately their satisfaction after surgery. The aim of this video is not to limit the doctor patient interaction (as all patients will still be granted their pre-allotted 30 minute visit with the physician regardless of their intervention allocation) but rather to augment the visit with additional educational information in an attempt to optimize the visit.

Objective:

A. Primary Aim(s):

• To determine if patients feel more prepared for surgery with addition of preoperative patient education video

B. Secondary Aim(s):

* To determine if addition of preoperative patient education video correlates with improved patient satisfaction after surgery
* To determine if patients' perception of time spent with healthcare team in preparation for surgery increases with addition of patient educational video
* To determine if actual patient-physician time spent counseling differs between groups
* To determine if patient preparedness is correlated with objective surgical outcomes
* To determine if patient preparedness is correlated with patient symptom improvement scores after surgery

Hypothesis:

The addition of a preoperative patient education video enhances patient preparedness for surgery, increases perception of the amount of time patients spend with healthcare team, and improves patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 scheduled to undergo either a laparoscopic or robotic-assisted sacrocolpopexy
* It is acceptable if concomitant procedures such as suburethral slings or additional vaginal repairs are planned
* English speaking
* Willing and able to provide written and informed consent

Exclusion Criteria:

* Women <18
* Not scheduled to undergo either a laparoscopic or robotic-assisted sacrocolpopexy
* Non-English speaking
* Unable or unwilling to provide written and informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
patients' preparedness for surgery | prior to surgery (baseline)
  patients' feelings of preparedness for surgery as determined by a preoperative patient preparedness questionnaire for pelvic surgery
Patient preparedness for surgery | 2 week postop visit
  patients' feelings of preparedness for surgery as determined by a postoperative patient preparedness questionnaire for pelvic surgery

SECONDARY OUTCOMES:
patient satisfaction | 2 weeks postop
  patient satisfaction as determined by completion of an adapted postoperative satisfaction questionnaire
perception of time | prior to surgery (baseline)
  patients' perception of time spent with healthcare team
Actual facetime spent | prior to surgery (baseline)
  Actual facetime spent between physician and patient during preoperative counseling session measured in minutes
QOL | 2 weeks postop
  Completion of validated condition specific QOL measures (ie. the Patient Global Impression of Improvement [PGI-I])
POPQ | 2 weeks postop
  Objective measures of success will be determined using the Pelvic organ prolapse quantification (POPQ to quantify prolapse)
Patient satisfaction | prior to surgery (baseline)
  patient satisfaction as determined by completion of an adapted preoperative satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Greene, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida Urogynecology clinic, Tampa, Florida, United States

REFERENCES:
- [Derived] Greene KA, Wyman AM, Scott LA, Hart S, Hoyte L, Bassaly R. Evaluation of patient preparedness for surgery: a randomized controlled trial. Am J Obstet Gynecol. 2017 Aug;217(2):179.e1-179.e7. doi: 10.1016/j.ajog.2017.04.017. Epub 2017 Apr 18. PMID 28431952